CLINICAL TRIAL: NCT01771380
Title: Measurement of the Free Fraction of 25-hydroxyvitamin D in Serum
Status: Completed | Type: Observational
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: Tromsø-Endo-2013-1
Record Dates: First submitted 2013-01-10; First posted 2013-01-18 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with impaired glucose tolerance

SUMMARY:
In the circulation 25-hydroxyvitaminD (25(OH)D) is bound to the vitamin D binding protein (DBP) and albumin. According to the free hormone hypothesis, it is, however, the free fraction that is biologically active. Polymorphisms in DBP are related to the serum level of 25(OH)D. As these polymorphisms may also affect the binding affinities for 25(OH)D, the total serum 25(OH)D may not necessary reflect the free fraction. To test this hypothesis, we will calculate the free fraction of 25(OH)D by correction for DBP and albumin content, and also measure free 25(OH)D from equilibrium dialysis and ultra filtration. Furthermore, we will relate total serum 25(OH)D as well as the free and biologically active (free- albumin-bound) 25(OH)D to the well established vitamin D effect marker serum parathyroid hormone as well as to the RNA expression in peripheral blood to evaluate the biological importance of the free versus the total fraction of 25(OH)D. We will invite 300 subjects from an ongoing vitamin D supplementation study to participate in the study which will be one visit only and include collection of blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance
* living in the Tromsø area

Exclusion Criteria

* pregnancy
* serious illness

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with known impaired glucose tolerance
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Free fraction of 25(OH)D | 1 day

SECONDARY OUTCOMES:
DBP polymorphisms | 1 day

OTHER OUTCOMES:
RNA expression in peripheral blood | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tromsø, Tromsø, Tromsø, Norway